CLINICAL TRIAL: NCT01680146
Title: Impact of Fat Co-ingestion With Protein on the Post-prandial Anabolic Response in Elderly Men (Pro-Fat Study)
Brief Title: Impact of Fat Co-ingestion With Protein on the Post-prandial Anabolic Response in Elderly Men
Acronym: Pro-Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: METC 12-3-030
Record Dates: First submitted 2012-08-21; First posted 2012-09-07 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Caseins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRO (Active Comparator): Subjects will ingest 20 g of intrinsically labeled casein dissolved in water
  Interventions: Dietary Supplement: PRO
- PRO+FAT (Experimental): Subjects will ingest 20 g of intrinsically labeled casein plus 26.7 g of anhydrous milk fat dissolved in water
  Interventions: Dietary Supplement: PRO+FAT

INTERVENTIONS:
Dietary Supplement: PRO+FAT
  Other Names: 20 g of casein + 26.7 g Anhydrous Milk Fat
  Arms: PRO+FAT
Dietary Supplement: PRO
  Other Names: 20 g of casein
  Arms: PRO

SUMMARY:
Rationale: The progressive loss of skeletal muscle mass with aging, or sarcopenia, has a major impact on our healthcare system due to increased morbidity and greater need for hospitalization and/or institutionalization. One way to prevent skeletal muscle loss is to improve dietary intake of the elderly. It has already been shown that ingestion of dietary protein stimulates muscle protein synthesis and inhibits muscle protein breakdown, resulting in an overall positive net protein balance. However, the impact of fat (as part of the meal) on dietary protein-induced muscle protein synthesis remains largely unknown. Based on previous studies by other research groups, we hypothesize that fat further stimulates the muscle anabolic response to protein ingestion.

Objective: The primary objective of this study is to investigate the effect of a single meal-like amount of protein with or without fat on postprandial muscle protein synthesis rates in healthy elderly men. Furthermore, as a secondary objective, we will assess digestion and absorption kinetics.

Study design: double-blind randomized intervention study Study population: 24 healthy elderly men (55-85 y) Intervention: one group (n=12) will consume a test beverage of 350 mL containing 20 g of intrinsically labeled casein, and the other group (n=12) will consume a beverage of the same volume containing 20 g of casein plus 20 g of fat.

Main study parameters/endpoints: Primary endpoint: muscle protein synthesis rates. Secondary endpoint: digestion and absorption kinetics.

DETAILED DESCRIPTION:
The progressive loss of skeletal muscle mass with aging, or sarcopenia, has a major impact on our healthcare system due to increased morbidity and greater need for hospitalization and/or institutionalization. The age-related loss of skeletal muscle mass is facilitated by a combination of factors, which include a less than optimal diet and a sedentary lifestyle. These factors contribute to a disruption in the regulation of skeletal muscle protein turnover, leading to an imbalance between muscle protein synthesis (MPS) and degradation. One way to overcome this problem is to improve dietary intake of the elderly. It has been well established that nutrient intake greatly affects protein turnover in skeletal muscle tissue.

Ingestion of dietary protein stimulates MPS rates and inhibits muscle protein breakdown rates, resulting in an overall positive net protein balance in both the young and elderly. However, it is not clear what the impact is of co-ingestion of other macronutrients on digestion and absorption kinetics or MPS rates in the healthy young or the elderly. We have recently conducted a study to examine the impact of carbohydrate co-ingestion on postprandial MPS in the healthy young and old. Indeed, preliminary results show that carbohydrate co-ingestion stimulates protein synthesis.

Interestingly, very little is known about the impact of fat co-ingestion with protein on the stimulation of post-prandial MPS rates. What is noteworthy is that Elliot et al. investigated the effect of whole milk ingestion on net muscle protein balance after resistance exercise using an arteriovenous balance approach. Ingestion of whole milk (containing 50 en% fats) stimulated the post-exercise net uptake of phenylalanine and threonine to a greater extent than ingestion of fat-free milk (containing 6 en% fat). Although, amino acid uptake is indicative of 'muscle anabolism', it is not a direct measure of MPS so no firm conclusions can be deduce from this work. Furthermore, milk also contains a certain amount of carbohydrates (fat-free milk 55 en% and whole milk 30 en%), which does not allow for direct assessment of fat co-ingestion per se.

Certainly, other studies have investigated the effect of long term fatty acid intake, using direct incorporation methods, on the MPS rates. For example, long term omega-3 polyunsaturated fatty acid (n-3 PUFA) supplementation increased feeding-mediated MPS rates in young, middle-aged, and older adults. The mechanism(s) underpinning the enhanced effect of n-3 PUFA supplementation on post-prandial MPS rates to dietary protein are not well defined. It has been speculated that the enhanced feeding-effect of n-3 PUFA on postprandial MPS rates is due to remodeling of the sarcolemma to include a greater n-3 PUFA content, and ultimately enhances insulin's action on muscle protein metabolism. This is clearly a long term effect, but what about the acute effects of fat co-ingestion on postprandial MPS rates? Katsanos et al. found that elevated plasma fatty acid concentrations did not interfere with the post-prandial stimulation of MPS. However, subjects ingested a single bolus of essential amino acids while receiving fatty acid infusion, which clearly does not reflect a 'real world' setting. In the end, there is reason to believe that the presence of fat in a meal further stimulates the muscle anabolic response to meal ingestion. However, fat intake may also modulate gastric emptying and dietary protein digestion and absorption kinetics. To date, the acute (not long-term supplementation) impact of fat in a meal on post-prandial muscle protein anabolism and digestion and absorption kinetics remains completely unexplored, and thus we can only speculate on the impact that fat co-ingestion has on postprandial MPS rates.

In the present study we will investigate the effect of a single meal-like amount of protein with or without fat on postprandial MPS in healthy elderly men. Furthermore, we will assess digestion and absorption kinetics. The use of intrinsically labeled casein will allows us determine de novo MPS from amino acids that come available through the test beverage.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Age between 55 and 85
* BMI < 30 kg/m2

Exclusion Criteria:

* Glucose intolerance
* Milk and/or fat intolerance
* Smoking
* Diagnosed GI tract diseases
* Arthritic conditions
* A history of neuromuscular problems
* Any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications).
* Use of anticoagulants
* Participation in exercise program
* Hypertension, high blood pressure that is above 140/90 mmHg.

Ages: 55 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
muscle protein synthesis (MPS) rates | 1 day
  The main study endpoint is muscle protein synthesis (MPS) rates. In order to determine the MPS, the following parameters will be measured:
  * Muscle protein-bound L-[1-13C]-phenylalanine, L-[ring-2H5]-phenylalanine, and L-[1-13C]-leucine enrichment (expressed as MPE)
  * Plasma L-[1-13C]-phenylalanine and L-[1-13C]-KIC enrichment (expressed as MPE)
  * Muscle free (intracellular) L-[1-13C]-phenylalanine enrichment (expressed as MPE)

SECONDARY OUTCOMES:
protein digestion and absorption kinetics | 1 day
  Secondary endpoints include protein digestion and absorption kinetics. Therefore, the following parameters will be measured:
  * Plasma phenylalanine, tyrosine, and leucine concentration (expressed as μmol/L)
  * Plasma enrichments of:
    * L-[1-13C]-phenylalanine
    * L-[1-13C]-tyrosine
    * L-[1-13C]-leucine
    * L-[ring-2H5]-phenylalanine
    * L-[ring-2H4]-tyrosine
    * L-[ring-2H2]-tyrosine
whole-body protein metabolism | 1 day
  Secondary endpoints include whole-body protein metabolism, which will be calculated based on protein digestion and absorption kinetics.
Glucose concentrations | 1 day
  During the experimental trial, we will measure glucose concentrations in the obtained plasma samples.
Insulin concentrations | 1 day
  During the experimental trial, we will measure insulin concentrations in the obtained plasma samples.

CONTACTS AND LOCATIONS:
Overall Officials: Luc JC van Loon, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Gorissen SHM, Trommelen J, Kouw IWK, Holwerda AM, Pennings B, Groen BBL, Wall BT, Churchward-Venne TA, Horstman AMH, Koopman R, Burd NA, Fuchs CJ, Dirks ML, Res PT, Senden JMG, Steijns JMJM, de Groot LCPGM, Verdijk LB, van Loon LJC. Protein Type, Protein Dose, and Age Modulate Dietary Protein Digestion and Phenylalanine Absorption Kinetics and Plasma Phenylalanine Availability in Humans. J Nutr. 2020 Aug 1;150(8):2041-2050. doi: 10.1093/jn/nxaa024. PMID 32069356
- [Derived] Gorissen SHM, Burd NA, Kramer IF, van Kranenburg J, Gijsen AP, Rooyackers O, van Loon LJC. Co-ingesting milk fat with micellar casein does not affect postprandial protein handling in healthy older men. Clin Nutr. 2017 Apr;36(2):429-437. doi: 10.1016/j.clnu.2015.12.011. Epub 2015 Dec 24. PMID 26774526
- See also: Research group website — http://www.m3-research.nl